CLINICAL TRIAL: NCT00006472
Title: Esophageal Cancer: A Phase II Study of Paclitaxel, Carboplatin and 5-Fluorouracil With Simultaneous Radiotherapy Followed by Surgical Resection
Brief Title: Combination Chemotherapy Plus Radiation Therapy Followed By Surgery in Treating Patients With Stage I, Stage II, or Stage III Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068295; WHC-99692; NCI-V00-1633
Record Dates: First submitted 2000-11-06; First posted 2004-02-26 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2002-02

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Carboplatin; Fluorouracil; Paclitaxel; Radiotherapy

ARMS (1):
- Single arm study (Other): Taxol® (Paclitaxel), Carboplatin and 5-Fluorouracil with Simultaneous Radiotherapy Followed by Surgical Resection
  Interventions: Drug: carboplatin; Drug: fluorouracil; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Carboplatin AUC 6 days 1 and 22
  Other Names: paraplatin
Drug: fluorouracil — 5FU 225mg/m2 continuous infusion on days 1-42 during radiation
  Other Names: 5FU
Drug: paclitaxel — taxol
  Other Names: 200mg/m2 days 1 and 22
Procedure: conventional surgery
Radiation: radiation therapy — The initial fields should be treated AP:PA when possible to a dose of 4500 cGy in 180 cGy fractions

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving chemotherapy drugs and radiation therapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy given before surgery in treating patients who have stage I, stage II, or stage III esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the total response rate in patients with stage I, II, or III esophageal cancer treated with paclitaxel, carboplatin, and fluorouracil with concurrent radiotherapy followed by surgical resection. II. Determine the overall survival of these patients treated with this regimen. II. Determine the toxicity of this regimen in this patient population.

OUTLINE: Patients receive paclitaxel IV over 1 hour followed by carboplatin IV over 30 minutes on days 1 and 22, and fluorouracil IV continuously on days 1-42. Patients undergo radiotherapy concurrently with chemotherapy daily 5 days a week for 5 weeks. Patients then undergo surgical resection within 3-5 weeks following completion of therapy. Patients are followed every 3 months for 6 months, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma or adenocarcinoma of the upper, middle, or lower third esophagus Stage I, II, or III disease Measurable disease No distant metastases Negative liver biopsy Negative bone scan unless due to benign disease No tracheobronchial involvement No vocal cord paralysis No phrenic nerve involvement No celiac axis lymph node involvement unless due to primary cancer at gastroesophageal junction No evidence of disseminated cancer

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT/SGPT no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No uncontrolled or severe cardiovascular disease No congestive heart failure No myocardial infarction within the past 6 months No severe or uncontrolled hypertension (systolic greater than 150 mmHg and diastolic greater than 100 mmHg) Pulmonary: FEV1/FVC at least 75% predicted Arterial blood saturation at least 92% Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other malignancy except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix No other serious medical illness that would limit survival to fewer than 2 years No active uncontrolled bacterial, viral, or fungal infection No active uncontrolled duodenal ulcer No psychiatric disorder that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior chest radiotherapy Surgery: No prior surgical resection of tumor Other: No prior therapy for esophageal cancer

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2000-01; Primary Completion 2001-11-15 (Actual); Study Completion 2002-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Perry, MD, Study Chair — Medstar Health Research Institute
Locations (6):
- United States (6):
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Union Memorial Hospital, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Good Samaritan Hospital of Maryland, Baltimore, Maryland